CLINICAL TRIAL: NCT07302412
Title: The Effect of Paternal Touch on Sucking Performance, Comfort, and Glucose Levels in Newborns at Risk for Hypoglycemia During the First Hours of Life
Brief Title: Effect of Paternal Touch on Sucking Performance, Comfort, and Glucose Levels in Newborns at Risk for Hypoglycemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Semra Küçük, Lecturer, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2025/18
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Infant, Newborn
Keywords: Gentle Human Touch; Paternal Touch; Newborn Feeding Performance; Comfort; Infant,; Blood Glucose; Newborn

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment randomized controlled design. Eligible newborns are randomly allocated to either the intervention group, in which paternal Gentle Human Touch is applied hourly for 15 minutes over the first 6 postnatal hours, or the control group, which receives routine care only. Randomization is performed using block randomization to ensure balanced allocation. Both groups are assessed in parallel at baseline, during the first breastfeeding session, and at the 2nd and 6th hours for feeding performance (LATCH), comfort level (COMFORTneo), and blood glucose values. No crossover between groups occurs.
Masking Description: Two independent assessors evaluate newborn feeding performance (LATCH) and comfort (COMFORTneo). The secondary assessor is blinded to group allocation and does not participate in the intervention. Both assessors perform evaluations independently and are blinded to each other's measurements to minimize observer bias."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentle Human Touch Group (Experimental): The father will apply Gentle Human Touch (GHT) following a structured protocol. After the newborn's routine care and baseline comfort assessment are completed in the baby care room, the first GHT session will begin. The father will place warm, steady hands on the newborn's head and pelvis, providing gentle, still touch for 15 minutes. This intervention will be repeated once every hour for the first 6 hours of life (a total of 6 sessions). No other additional interventions will be applied. Feeding performance, comfort level, and blood glucose values will be assessed according to the study protocol.
  Interventions: Procedure: Gentle Human Touch
- Standard Care Group (Other): Newborns in this group will receive routine clinical care only. No Gentle Human Touch or any other additional intervention will be applied. Baseline comfort assessment will be performed after routine care, and feeding performance, comfort level, and blood glucose values will be evaluated at the same time points as in the intervention group.
  Interventions: Other: Standard Care Group

INTERVENTIONS:
Procedure: Gentle Human Touch — The father will apply Gentle Human Touch (GHT) following a structured protocol. After the newborn's routine care and baseline comfort assessment are completed in the baby care room, the first GHT session will begin. The father will place warm, steady hands on the newborn's head and pelvis, providing gentle, still touch for 15 minutes. This intervention will be repeated once every hour for the first 6 hours of life (a total of 6 sessions). No other additional interventions will be applied. Feeding performance, comfort level, and blood glucose values will be assessed according to the study protocol.
  Arms: Gentle Human Touch Group
Other: Standard Care Group — Newborns in this group will receive routine clinical care only. No Gentle Human Touch or any other additional intervention will be applied. Baseline comfort assessment will be performed after routine care, and feeding performance, comfort level, and blood glucose values will be evaluated at the same time points as in the intervention group.
  Arms: Standard Care Group

SUMMARY:
This randomized controlled trial aims to examine the effects of Gentle Human Touch applied by fathers during the first hours of life on sucking performance, comfort level, and blood glucose values in newborns at risk for hypoglycemia. Eligible newborns will be randomly assigned to intervention and control groups.

After the newborn is taken to the baby care room and routine care procedures are completed, comfort level will be assessed by the primary nurse and an independent second observer using the Neonatal Comfort and Behavior Scale (NCBS). In the intervention group, the first Gentle Human Touch application will begin after routine care and the initial comfort assessment are completed. Sucking performance will be assessed during the first breastfeeding session by the primary nurse and an independent observer using the LATCH Breastfeeding Assessment Tool.

In the intervention group, fathers will administer 15-minute Gentle Human Touch sessions every hour for six hours according to a structured protocol. In the control group, routine care will be provided without any additional touch.

In both the intervention and control groups, blood glucose levels will be measured at the 2nd hour according to clinical protocols. At the 6th hour, the newborn's comfort level (NCBS), sucking performance (LATCH), and blood glucose level will be reassessed and recorded.

This study aims to determine whether early paternal touch supports glucose stability, improves sucking performance, and enhances comfort in newborns at risk for hypoglycemia, and to contribute to the development of family-centered, non-invasive care practices in neonatal settings.

DETAILED DESCRIPTION:
Neonatal hypoglycemia is one of the most common metabolic problems in the neonatal period and is particularly prevalent among infants with specific perinatal risk factors. Approximately one-third of newborns are considered at risk for hypoglycemia, and a substantial proportion develop low blood glucose values within the first 24-48 hours of life. Because failure to promptly recognize and treat hypoglycemia may lead to neurological injury, implementing interventions that support physiological stability during the first hours of life is critically important in at-risk newborns. Early skin-to-skin contact and initiation of breastfeeding contribute to the maintenance of glucose regulation and physiological stability; however, research examining the effects of structured paternal touch (Gentle Human Touch) in newborns at risk for hypoglycemia is extremely limited.

Gentle Human Touch (GHT) is a non-invasive intervention applied by healthcare professionals or parents, consisting of steady, warm, light hand placement on specific areas of the infant's body. Studies conducted in preterm and term infants have reported that GHT may reduce stress responses, support behavioral organization, and positively affect physiological parameters such as heart rate and oxygen saturation. Nevertheless, no studies have specifically examined the impact of paternal gentle touch on feeding performance, comfort, and glucose regulation in newborns. This research will be one of the first to evaluate whether paternal GHT improves early physiological and behavioral outcomes in newborns at risk for hypoglycemia.

The primary aim of this study is to determine the effects of paternal Gentle Human Touch applied during the first hours of life on sucking performance, comfort level, and blood glucose values in newborns. The null hypothesis states that paternal GHT has no effect on these outcomes, whereas the alternative hypothesis proposes that the intervention will improve sucking performance, increase comfort, and support glucose stability.

This single-center, randomized controlled experimental study will be conducted in the baby care room of Acibadem Mehmet Ali Aydinlar University Atakent Hospital. The study population consists of all newborns followed in the baby care room who are identified as being at risk for hypoglycemia. The sample will include newborns who meet the inclusion criteria and whose parents provide written informed consent. Based on a power analysis conducted using G*Power, with an effect size of 0.57, a 95% confidence level, and 80% power, a minimum of 49 newborns per group is required, resulting in a total sample size of 98.

Risk for hypoglycemia will be evaluated based on clinical factors including maternal diabetes, preeclampsia, pregnancy-induced hypertension, use of beta-blockers or other medications associated with neonatal hypoglycemia, prematurity, SGA/LGA status, intrauterine growth restriction, asphyxia, hypoxia, sepsis, polycythemia, hypothermia, metabolic or endocrine disorders, antepartum glucose administration, intravenous indomethacin use, and similar risk conditions. Newborns with major congenital anomalies or genetic syndromes, as well as those who develop hypoglycemia requiring treatment during the study period, will be excluded.

Randomization will be performed using a block randomization method with blocks of four, ensuring balanced allocation between the intervention and control groups throughout data collection. Newborns will be assigned sequentially according to the pre-generated randomization list.

Data will be collected using three main instruments: (1) the Neonatal Information Form, which records antenatal, birth, and postnatal characteristics; (2) the LATCH Breastfeeding Assessment Tool, which evaluates feeding performance across five domains; and (3) the Neonatal Comfort and Behavior Scale (NCBS/COMFORTneo), which assesses behavioral and physiological comfort. Permissions for scale use have been obtained.

After birth, the newborn is transferred to the baby care room, where routine assessments (physical examination, respiratory evaluation, temperature regulation) are completed. Once these procedures are finished, the newborn's baseline comfort level will be assessed by the primary nurse and an independent observer using the NCBS. In the intervention group, the first Gentle Human Touch session will begin immediately after this initial comfort assessment. Fathers will receive verbal instruction and illustrated training materials explaining the protocol (hand placement, pressure, duration) before the first session.

According to the GHT protocol, the father washes his hands and warms them to approximately 34°C. In a quiet, low-stimulus environment, he places one hand gently on the infant's head and the other on the pelvic region, maintaining steady touch without stroking for 15 minutes. This procedure will be repeated once every hour for the first six hours after birth, totaling six sessions. In the control group, newborns will receive routine care without any additional touch.

When the mother is clinically stable, the newborn will be brought for the first breastfeeding session. During this feeding, sucking performance will be evaluated by the primary nurse and the independent observer using the LATCH scale. Blood glucose levels will be measured at the 2nd hour of life in accordance with routine clinical protocols for at-risk infants.

At the 6th hour, after the final GHT session in the intervention group, the newborn's comfort level (NCBS), sucking performance (LATCH), and blood glucose value will be reassessed and recorded in both groups.

Ethical approval has been obtained from the Acibadem Mehmet Ali Aydinlar University Medical Research Evaluation Board (ATADEK). Written informed consent will be obtained from parents before participation. The intervention is entirely non-invasive and consists only of gentle, steady paternal touch; therefore, it poses minimal risk. Blood glucose measurements are part of routine clinical care and no additional sampling will be performed for research purposes. Any infant who develops hypoglycemia requiring treatment will be managed per institutional protocol and removed from the study.

The findings of this study are expected to contribute valuable evidence regarding the role of paternal touch in promoting physiological and behavioral stability in newborns at risk for hypoglycemia and to support the integration of low-cost, family-centered, non-invasive interventions into routine neonatal care practices.

ELIGIBILITY:
Inclusion Criteria:

* Newborns identified as being at risk for hypoglycemia (see study population).
* Newborns whose parents/legal guardians have provided written informed consent.
* Clinically stable newborns who have no contraindications to breastfeeding during the first 6 hours after birth.
* Newborns whose fathers are present during the first 6 hours after birth.

Exclusion Criteria:

* Newborns who develop hypoglycemia during the study period or who require initiation of hypoglycemia treatment.
* Newborns with congenital anomalies or a diagnosed genetic syndrome.

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-12-08 (Estimated); Study Completion 2027-12-08 (Estimated)

PRIMARY OUTCOMES:
Sucking Performance | During the first breastfeeding session and at the 6th hour
  Sucking performance will be assessed using the LATCH Breastfeeding Assessment Tool, which evaluates latch, audible swallowing, type of nipple, maternal comfort, and positioning. The total score ranges from 0 to 10, with higher scores indicating greater breastfeeding success, reflecting more effective sucking and better coordination. Assessments will be performed independently by the primary nurse and an independent second observer, who are blinded to each other's evaluations.
Newborn Comfort Level | After routine newborn care (baseline) and at the 6th hour
  Newborn comfort level will be assessed using the Newborn Comfort and Behavior Scale (COMFORTneo), which evaluates behavioral and physiological indicators of comfort. The total score ranges from 6 to 30, with higher scores indicating lower comfort and increased behavioral or physiological distress. After the newborn is taken to the baby care room and routine care is completed, assessments will be performed independently by the primary nurse and an independent second observer, who are blinded to each other's evaluations. A second assessment will be performed at the 6th hour.
Blood Glucose Level | At the 2nd hour and the 6th hour
  Blood glucose level will be measured using a standard glucometer according to routine clinical practice. The first measurement will be recorded at the 2nd hour, and the second measurement at the 6th hour. Importantly, blood glucose monitoring at these time points is part of the institution's routine protocol; therefore, no additional measurements are performed for research purposes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belpinar A, Yayan EH. Effect of Yakson touch and mother's voice on pain and comfort level during nasal CPAP application in Turkey: A randomized controlled study. Explore (NY). 2023 Sep-Oct;19(5):743-748. doi: 10.1016/j.explore.2023.02.010. Epub 2023 Feb 20. PMID 36872192
- [Background] Cobo MM, Moultrie F, Hauck AGV, Crankshaw D, Monk V, Hartley C, Evans Fry R, Robinson S, van der Vaart M, Baxter L, Adams E, Poorun R, Bhatt A, Slater R. Multicentre, randomised controlled trial to investigate the effects of parental touch on relieving acute procedural pain in neonates (Petal). BMJ Open. 2022 Jul 19;12(7):e061841. doi: 10.1136/bmjopen-2022-061841. PMID 36250332
- [Background] Kilinc D, Caglar S. The Effect of Mother's Gentle Human Touch on Preterm Neonate's Pain and Maternal Anxiety During Venipuncture in Turkiye. Res Nurs Health. 2025 Aug;48(4):487-496. doi: 10.1002/nur.22472. Epub 2025 May 20. PMID 40392177
- [Background] Sezer Efe Y, Erdem E, Caner N, Gunes T. The effect of gentle human touch on pain, comfort and physiological parameters in preterm infants during heel lancing. Complement Ther Clin Pract. 2022 Aug;48:101622. doi: 10.1016/j.ctcp.2022.101622. Epub 2022 Jun 22. PMID 35759976